CLINICAL TRIAL: NCT01299961
Title: Musculoskeletal Ultrasound as a Marker of Therapeutic Response to Abatacept in Rheumatoid Arthritis
Brief Title: Ultrasound Scores as Indication of Response to Subcutaneous Abatacept in Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Dr. Veena Ranganath, M.D., Assistant Clinical Professor, University of California, Los Angeles
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: UCLA Rheumatology RA 001; IND 111281 (Other: FDA)
Record Dates: First submitted 2011-02-18; First posted 2011-02-21 (Estimated); Results first posted 2015-01-30 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-05

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Subcutaneous Abatacept; Ultrasound
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subcutaneous Abatacept (Experimental): All subjects will receive an injection of 125 mg of abatacept once a week up to 12 months.
  Interventions: Drug: abatacept

INTERVENTIONS:
Drug: abatacept — 125 mg once a week up to 12 months.

SUMMARY:
Rheumatoid arthritis (RA) is a chronic inflammatory disease (a long-lasting disease causing pain and swelling) associated with significant health problems. It is a difficult disease to manage as the disease is often unpredictable. RA causes inflammation (swelling) of the joints that can cause joint damage, deformity, and progressive disability and impairment. It is estimated that 1% of the world's population suffers from this disease.

The purpose of this research study is to determine if a change in inflammation seen on the ultrasound is a good indicator of how subjects' rheumatoid arthritis is responding to treatment of subcutaneous abatacept at 3 weeks, 3 months, 6 months, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years old
2. Has a diagnosis of rheumatoid arthritis
3. Stable DMARDs for at least 1 month (methotrexate, leflunomide, hydroxychloroquine, or sulfasalazine)
4. Disease activity score DAS28/ESR > 3.2 or all must be met: TJC (tender joint count)>=4, SJC (swollen joint count)>=4
5. Must be able to understand information in the Informed Consent and comply with study requirements
6. Total ultrasound synovitis (inflammation of joint-lining membrane) power Doppler score >=1 for at least 2 joints and total synovitis score >=1 for at least 1 joint

Exclusion Criteria:

1. Current or prior use of biologic drugs (TNF inhibitors, IL-6 inhibitors, CD20 inhibitors, IL-1 inhibitors, etc.)
2. Pregnancy or breast feeding
3. Daily prednisone > 10mg (stable dose for at least 1 month)
4. Intra-articular steroid injection of the wrist or joints within last 2 months
5. History of a concomitant autoimmune disease such as lupus, psoriatic arthritis
6. History of cancer
7. Previous exposure to abatacept

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-03; Primary Completion 2013-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Veena K Ranganath, M.D., Principal Investigator — UCLA David Geffen School of Medicine, Division of Rheumatology
Locations (1):
- UCLA David Geffen School of Medicine, Division of Rheumatology, Los Angeles, California, United States

REFERENCES:
- [Derived] Charles-Schoeman C, Wang J, Shahbazian A, Wilhalme H, Brook J, Kaeley GS, Oganesian B, Ben-Artzi A, Elashoff DA, Ranganath VK. Power doppler ultrasound signal predicts abnormal HDL function in patients with rheumatoid arthritis. Rheumatol Int. 2023 Jun;43(6):1041-1053. doi: 10.1007/s00296-023-05285-7. Epub 2023 Feb 24. PMID 36828925

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 34 RA patients were recruited from the UCLA rheumatology clinics between September 2011 to February 2013. However, we had a total of 9 screen fails.
Pre-assignment Details: Patients enrolled in the study were required to have RA, on stable RA medications, and naive to abatacept.
Period: Overall Study
Arm/Group | Subcutaneous Abatacept
Started | 25
Completed | 19
Not Completed | 6
Not completed — Adverse Event | 3
Not completed — Lack of Efficacy | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Subcutaneous Abatacept
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] — This is a the average age of the cohort that started the mediation, Abatacept 125mg sq qwk.
  years | 52.6 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: 12 Month Change in 7-Joint Ultrasound (US) Inflammatory Score
Description: The 7-joint US inflammatory score includes the addition of synovial hypertrophy scores and power doppler scores.
Time Frame: baseline, 12 months
Population: Total of 19 patients completed 12 mos
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Subcutaneous Abatacept
Number analyzed (Participants) | 19
units on a scale | 11.4 (13.1)
Statistical Analysis 1: Comparison: Subcutaneous Abatacept; Most involved side: Synovitis (S), tenosynovitis (T), and power Doppler (PD) of wrist (dorsal (D), palmar (P), and ulnar (U)); S and T of MCP 2,3 (P, plus D for T); PD of the MCP joints (P and D); S and PD of PIP 2, 3 (P, plus D for PD); S and PD for MTP 2, 4 (D). S and PD graded from 0 to 3, and max individual scores are 27 and 39, respectively. T graded on 0-1 scale; max T score is 5. High score is worse. The 7-joint US score is sum of T, S, and PD scores. Change calculated baseline- month 12; Test type: Superiority or Other; p < 0.01, t-test, 2 sided; Mean Difference (Final Values) = 11.4, Standard Deviation 13.1

2. Secondary Outcome: 12 Month Change in Power Doppler Ultrasound (PDUS) Scores
Description: There were seven different joints in the hands and wrists evaluated to score the PDUS.
Time Frame: baseline, 12 months
Population: As stated previously
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Subcutaneous Abatacept
Number analyzed (Participants) | 19
units on a scale | 3.0 (3.7)
Statistical Analysis 1: Comparison: Subcutaneous Abatacept; 7 joints were scanned by power doppler ultra sound of the most affected side: wrist, MCP 2/3, PIP 2/3, and MTP 2/5. PDUS was scored semi-quantitatively on a scale of 0-3 (higher score is worse). The mean score of the 2-3 views obtained for each joint was added across all 7 joints, and the total PDUS (range 0-21) scores were calculated. The change from baseline to 12 months is calculated as the baseline PDUS minus 12 month PDUS; Test type: Superiority or Other; p < 0.01, t-test, 2 sided; Mean Difference (Final Values) = 3.0, Standard Deviation 3.7

3. Secondary Outcome: 12 Month Change in Gray-scale Ultrasound (GSUS)
Description: There were seven different joints in the hands and wrists evaluated to score the GSUS.
Time Frame: baseline, 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Subcutaneous Abatacept
Number analyzed (Participants) | 19
units on a scale | 1.2 (3.7)
Statistical Analysis 1: Comparison: Subcutaneous Abatacept; 7 joints were scanned by grey-scale ultra sound of the most affected side: wrist, MCP 2/3, PIP 2/3, and MTP 2/5. GSUS was scored semi-quantitatively on a scale of 0-3 (higher score is worse). The mean score of the 2-3 views obtained for each joint was added across all 7 joints, and the total GSUS (range 0-21) scores were calculated. The change from baseline to 12 months is calculated as the baseline GSUS minus 12 month GSUS; Test type: Superiority or Other; p = 0.19, t-test, 2 sided; Mean Difference (Final Values) = 1.2, Standard Deviation 3.7

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Subcutaneous Abatacept
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

LIMITATIONS AND CAVEATS:
This is a very small open-label study of 25 patients on a FDA approved drug, where efficacy (by standard validated measures) and safety were not the primary end points.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No